CLINICAL TRIAL: NCT06324149
Title: Age-related Conditions in the Context of Multimorbidity and Frailty: Relative Weight of Frailty in Determining the Course and Outcomes of Different Chronic Diseases and Viceversa
Acronym: AGE-IT-FRAILTY
Status: Recruiting | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Rovere Querini Patrizia, Professor, IRCCS San Raffaele
Other Study IDs: AGE-IT-FRAILTY
Record Dates: First submitted 2024-03-05; First posted 2024-03-21 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Frailty; Sarcopenia
MeSH Terms: conditions — Frailty; Sarcopenia | interventions — Blood Specimen Collection; Electrocardiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — FGF21, GDF15, Nfl, sRAGE, HMGB1
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- older volunteers: 1250 individuals of the FRASNET study (original promoter of the study Ospedale San Raffaele, Principal Investigator Professor Paolo Manunta): older volunteers who were either robust or frail at the evaluations performed in 2016-2017)
  * completion of scales and questionnaires
  * venous blood sampling
  * muscle ultrasound
  * cardiac ultrasound
  * electrocardiogram
  * bioelectrical impedance analysis
  Interventions: Diagnostic Test: completion of scales and questionnaires; venous blood sampling; muscle ultrasound; cardiac ultrasound; electrocardiogram; bioelectrical impedance analysis
- neurology patients: 720 patients suffering from cognitive impairment and clinically followed at the Neurology Department of the San Raffaele Hospital (UniSR Prof Agosta)
  * completion of scales and questionnaires
  * venous blood sampling
  * muscle ultrasound
  * cardiac ultrasound
  * electrocardiogram
  * bioelectrical impedance analysis
  Interventions: Diagnostic Test: completion of scales and questionnaires; venous blood sampling; muscle ultrasound; cardiac ultrasound; electrocardiogram; bioelectrical impedance analysis

INTERVENTIONS:
Diagnostic Test: completion of scales and questionnaires; venous blood sampling; muscle ultrasound; cardiac ultrasound; electrocardiogram; bioelectrical impedance analysis — The sub-investigator performs a multidimentional geriatric evaluation

SUMMARY:
Observational study. Participants of the FRASNET study (9th March 2017, Protocol No. 24/INT/2017) who were evaluated in 2016 and 2017 will be contacted to be re-evaluated with multidimensional visits as part of the present study in order to assess trajectories and biomarkers of frailty and sarcopenia. Moreover, are going to evaluate with the same multidimensional visits patients with mild cognitive impairment and dementia followed up at the Neurologic Unit of the San Raffaele Hospital.

ELIGIBILITY:
Inclusion Criteria:

* Having participated in the FRASNET study or being a patient with mild cognitive impairment or dementia followed up at the Neurologic Unit of the San Raffaele Hospital
* Ability to sign written informed consent
* > 18 years old

Exclusion Criteria:

* Life expectancy < 6 months
* Unwillingness to participate in the study
* Unstable clinical disease(for ex. serious acute pathologies)

Ages: 18 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: * 1250 individuals of the FRASNET study (original promoter of the study Ospedale San Raffaele, Principal Investigator Professor Paolo Manunta): older volunteers who were either robust or frail at the evaluations performed in 2016-2017 )
  * 720 patients suffering from cognitive impairment and clinically followed at the Neurology Department of the San Raffaele Hospital (UniSR Prof Agosta)
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-03-07 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
identify new molecular markers of frailty and sarcopenia | febbrary 2026
  To identify new molecular markers of frailty and sarcopenia in elderly volunteers and patients suffering from mild cognitive impairment and dementia assay of biomarkers (HMGB1, sRAGE, FGF21, GFD15 and neurofilaments)

SECONDARY OUTCOMES:
evaluate the ability of new markers for frailty, sarcopenia, cognitive impairment | april 2026
  To evaluate the ability of new markers (identified through the analysis of biobanked blood samples) to predict individual trajectories of frailty, sarcopenia, cognitive impairment and clinical outcomes assay of biomarkers (HMGB1, sRAGE, FGF21, GFD15 and neurofilaments)

CONTACTS AND LOCATIONS:
Locations (1):
- San Raffaele Hospital, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided